CLINICAL TRIAL: NCT04264260
Title: Evaluation the Palliative Effects of Colchicine on Primary Hepatic Malignant Tumors Unable to Receive Curative Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Zu-Yau Lin, professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20190152
Record Dates: First submitted 2020-02-02; First posted 2020-02-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma Stage IIIB; Cholangiocarcinoma, Intrahepatic; Cholangiocarcinoma; With Hepatocellular Carcinoma; Hepatocellular Carcinoma Stage IV
Keywords: hepatocellular carcinoma; Cholangiocarcinoma; primary hepatic malignancy; palliative treatment; colchicine
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Liver Neoplasms | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: open labeled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- colchicine group (Experimental): The participants will receive colchicine starting from 2 tablets after meal twice per day (total 2 mg). The dose will be adjusted ranging from total minimum 1.5 mg to maximum 3 mg per day based on the condition and tolerance of the participant. One cycle of treatment is defined as 4 days treatment and 3 days off. The participants will receive repeated cycles till the participants quit the trial.
  Interventions: Drug: Colchicine Tablets

INTERVENTIONS:
Drug: Colchicine Tablets — three times or two times per day after meal with the daily total dose ranging from 1.5 to 3 mg

SUMMARY:
This trial is to evaluate the palliative effects of colchicine on primary hepatic malignancy using the Department of Health R.O.C. approved doses and methods of administration. Colchicine will be started from 2 tablets after meal twice per day (total 2 mg), adjust the dose ranging from total minimum 1.5 mg to maximum 3 mg per day based on the condition and tolerance of the participant. One cycle of treatment is defined as 4 days treatment and 3 days off. The participants will receive repeated treatment cycles till the participants quit the trial. The control group will be originated from review of (1) patients treated by members of this research team with the same condition as the trial selected participants but not included in the trial, (2) patients with same condition as the trial selected participants reported in the literatures. The primary objective is to evaluate the palliative effects of colchicine on primary hepatic malignancy unable to receive curative treatment. The primary end point is survival of the participant. The Secondary objective is to evaluate the safety of patients treated by colchicine and the secondary end point is the side effects of colchicine.

DETAILED DESCRIPTION:
Study procedures

1. Written informed consent before study specific procedures are undertaken. The investigators will explain the contents of the trial especially the information about the possible side effects, other alternative treatment and the right to withdraw based on the participant own willing to the candidates. Patient can choose to sign or not to sign the inform consent based on his/her own decision after completely understanding the investigators explanation.
2. The process of the experiment

Start to receive colchicine:

Participant will start to receive colchicine starting from 2 tablets after meal twice per day (total 2 mg).

Adjustment the dosage of colchicine during study: based on the following steps:

2 tablets-2 tablets-2 tablets (three times per day, after meal, total 3 mg, maximum dose)<-> 2 tablets -1 tablet -2 tablets (three times per day, after meal, total 2.5 mg)<->2 tablets -2 tablets (twice per day, after meal, 2 mg, starting dose)<->1 tablet -1 tablet -1 tablet (three times per day, after meal, 1.5 mg, minimum dose)

1. The colchicine dosage will be changed when the hepatic reserved function of the participant changes to Child score 8-9 points according to the following rules.

   1. 1 tablet after meal three times per day with total dose of 1.5 mg; continue 4 days and stop for 3 days (1 cycle)
   2. If the hepatic reserved function of the participant returns to Child score < 8 points, the dosage changes to starting dose.
   3. If the hepatic reserved function of the participant changes to Child score > 9 points, colchicine will be stopped and participant receives regular follow-up only.
2. If participant suffers from severe diarrhea, colchicine will be temporarily stopped. When the symptom of diarrhea subsides, colchicine will be given again according to the above steps of dose adjustment.
3. If the participant has one of the following conditions, colchicine will be temporarily stopped. When the condition of the participant improves, colchicine will be given again after the judgment from the doctor of the research team. For participants unable to receive colchicine again, they will receive regular follow-up only.

   1. . There are life-threatening hemorrhage including gastrointestinal hemorrhage and hemorrhage from other vital organs such as lungs or brain.
   2. . There are life-threatening bacterial, fungal or viral infection (not included hepatitis B and C virus).
   3. . Patient has serum creatinine level > 1.5 mg/dL.
   4. . Patient has white blood cell count < 1500/µL, platelet count < 30000/µL or hemoglobin < 9.0 gm/dL after medication.
   5. . The research team decides that the participant is not suitable to continue the study caused by abnormality of any vital organ or severe side effects caused by the study.
4. Colchicine will be temporarily stopped before non-curative operative resection of tumor or transcatheter arterial chemoembolization until participant has body temperature < 38 ℃, same hepatic reserved function as before, and serum creatinine level < 1.5 mg/dL.
5. no need to stop colchicine during irradiation therapy, pure ethanol injection or local radiofrequency abrasion
6. Colchicine needs to be temporarily reduced to half of the original dose when the participant will temporarily take P-Glycoprotein inhibitor or strong Cytochrome P450 3A4 inhibitor.

The conditions for the participant to withdraw or terminate the trial:

1. Participant suffers from systemic itching, nausea, vomiting, abdominal pain, fever, or skin rash after colchicine administration.
2. Participant is unable to tolerate 1.5 mg total daily dose of colchicine for at least 4 cycles. This does not include temporarily reduce dose to total 1 mg during temporarily application of P-Glycoprotein inhibitor or strong Cytochrome P450 3A4 inhibitor.

Follow-up procedures and items for the participants to co-operate:

All participants will be followed according to the guide line of the National Health Council and the clinical practice in the treatment of hepatic malignancy. Ultrasonography, contrasted-enhanced computed tomography or magnetic resonance imaging will be performed within every 3 to 4 months. Chest x-ray and whole body bone scan will be followed based on the condition of the participants. Serum alpha-fetoprotein or CA19-9 will be determined within 3 months in participants with abnormal original levels. The complete blood count, hepatic and renal function will be determined at least one session every month. The participants are asked to visit investigators' outpatient clinic at least one session every month.

Concomitant treatment:

1. Permitted:

   non-curative operative resection of the tumor, local abrasion therapy, local irradiation therapy, transcatheter arterial chemoembolization, target therapy, immunotherapy
2. Prohibited:

systemic chemotherapy, other clinical trial testing drugs, Chinese traditional medicine, herb drugs

Statistical analysis

1.Statistical Method for Efficacy / Safety measurements: (A) Survival analysis for efficacy: (log-rank test and median survival)

* colchicine combined with other therapy is better than other therapy without target drug or immunotherapy
* colchicine combined with other therapy is not inferior than target drug or immunotherapy combined with other therapy (B) Safety measurements The safety assessment is presented in a narrative statistical manner for the collection of participants' severe adverse events and adverse events.

ELIGIBILITY:
Inclusion Criteria:

(A). Primary hepatic malignancy including hepatocellular carcinoma, intrahepatic cholangiocarcinoma, hepatocellular-cholangiocarcinoma, poorly differentiated or undifferentiated primary hepatic malignancy.

1. Diagnosis of hepatocellular carcinoma: Patient has at least one of the following criteria: (1) positive for hepatocellular carcinoma evidenced by cytology or pathology, (2) serum alpha-fetoprotein level > 400 ng/mL and has evidence of hepatocellular carcinoma on contrast-enhanced computed tomography or magnetic resonance imaging.
2. Diagnosis of intrahepatic cholangiocarcinoma: Patient has at least one of the following criteria: (1) evidenced by cytology or pathology, (2) serum CA19-9 level > 10 times of normal upper limit and has evidence on contrast-enhanced computed tomography or magnetic resonance imaging, and no evidence of extrahepatic original malignancy.
3. Diagnosis of hepatocellular-cholangiocarcinoma: concomitantly fit at least one of the items described in (a) and (b)
4. Diagnosis of poorly differentiated or undifferentiated primary hepatic malignancy: Patient fits all of the following criteria: (1) evidenced of malignancy other than hepatocellular carcinoma, intrahepatic cholangiocarcinoma or hepatocellular-cholangiocarcinoma by cytology or pathology, (2) no evidence of extrahepatic original malignancy

(B). Primary hepatic malignant tumors unable to receive curative treatment indicate that the malignancy can not be completely eliminated by operative resection, liver transplantation or local abrasion therapy. Patient also needs to fit at least one of the following criteria: (1) evidence of distant metastasis or large vessels (intrahepatic first branch portal vein, portal main trunk, major hepatic vein or inferior vena cava) invasion, (2) unable to be controlled by transcatheter arterial chemoembolization including appearance of new rather than incompletely treated nodules within 3 months of chemoembolization, or chemoembolization fails

(C). The performance status of the patient based on the Eastern Cooperative Oncology Group (ECOG) belongs to 0 or 1 and the calculated Child score is below 8 points.

Exclusion Criteria:

1. . life-threatening hemorrhage at the present time
2. . life-threatening bacterial, fungal or viral infection (not included hepatitis B and C virus) at the present time
3. . extrahepatic original malignancy unable to be controlled
4. . serum creatinine level > 1.5 mg/dL.
5. . Patient must receive long-term statin or fibrates drugs. The doses of these medications can not be altered.
6. . Patient has white blood cell count < 1500/µL, platelet count < 30000/µL or hemoglobin < 9.0 gm/dL after medication.
7. . Pregnant woman or plan to be a pregnant woman
8. . allergy to colchicine or has history of severe side effects caused by colchicine
9. . Patient has received systemic chemotherapy within 2 months before enrollment or plans to receive systemic chemotherapy in the future.
10. . Patient is under or plans to receive other clinical trial testing drug.
11. . Patient has severe malfunction of vital organs and can not participate in this study justified by the member of the research team.
12. . Patient is under or plans to receive Chinese traditional medicine or herb drugs.
13. . Patient is under or plans to receive hospice care.
14. . Patient took other clinical trial testing drug within 3 months before enrollment.
15. . Patient can not quit drug abuse or heavy alcohol drinking.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
survival | through study completion, an average of 31 months
  The overall survival of the participants

SECONDARY OUTCOMES:
serious adverse effect | through study completion, an average of 31 months
  The events of serious adverse effect occurred during the study

CONTACTS AND LOCATIONS:
Overall Officials: Zu Y Lin, MD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arrieta O, Rodriguez-Diaz JL, Rosas-Camargo V, Morales-Espinosa D, Ponce de Leon S, Kershenobich D, Leon-Rodriguez E. Colchicine delays the development of hepatocellular carcinoma in patients with hepatitis virus-related liver cirrhosis. Cancer. 2006 Oct 15;107(8):1852-8. doi: 10.1002/cncr.22198. PMID 16967451
- [Background] Finkelstein Y, Aks SE, Hutson JR, Juurlink DN, Nguyen P, Dubnov-Raz G, Pollak U, Koren G, Bentur Y. Colchicine poisoning: the dark side of an ancient drug. Clin Toxicol (Phila). 2010 Jun;48(5):407-14. doi: 10.3109/15563650.2010.495348. PMID 20586571
- [Background] Imazio M, Bobbio M, Cecchi E, Demarie D, Demichelis B, Pomari F, Moratti M, Gaschino G, Giammaria M, Ghisio A, Belli R, Trinchero R. Colchicine in addition to conventional therapy for acute pericarditis: results of the COlchicine for acute PEricarditis (COPE) trial. Circulation. 2005 Sep 27;112(13):2012-6. doi: 10.1161/CIRCULATIONAHA.105.542738. PMID 16186437
- [Background] Kallinich T, Haffner D, Niehues T, Huss K, Lainka E, Neudorf U, Schaefer C, Stojanov S, Timmann C, Keitzer R, Ozdogan H, Ozen S. Colchicine use in children and adolescents with familial Mediterranean fever: literature review and consensus statement. Pediatrics. 2007 Feb;119(2):e474-83. doi: 10.1542/peds.2006-1434. Epub 2007 Jan 22. PMID 17242135
- [Background] Leighton JA, Bay MK, Maldonado AL, Schenker S, Speeg KV. Colchicine clearance is impaired in alcoholic cirrhosis. Hepatology. 1991 Dec;14(6):1013-5. PMID 1959847
- [Background] Rochdi M, Sabouraud A, Girre C, Venet R, Scherrmann JM. Pharmacokinetics and absolute bioavailability of colchicine after i.v. and oral administration in healthy human volunteers and elderly subjects. Eur J Clin Pharmacol. 1994;46(4):351-4. doi: 10.1007/BF00194404. PMID 7957521
- [Background] Ferron GM, Rochdi M, Jusko WJ, Scherrmann JM. Oral absorption characteristics and pharmacokinetics of colchicine in healthy volunteers after single and multiple doses. J Clin Pharmacol. 1996 Oct;36(10):874-83. doi: 10.1002/j.1552-4604.1996.tb04753.x. PMID 8930773
- [Background] Terkeltaub RA, Furst DE, Bennett K, Kook KA, Crockett RS, Davis MW. High versus low dosing of oral colchicine for early acute gout flare: Twenty-four-hour outcome of the first multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-comparison colchicine study. Arthritis Rheum. 2010 Apr;62(4):1060-8. doi: 10.1002/art.27327. PMID 20131255
- [Background] Lin ZY, Wu CC, Chuang YH, Chuang WL. Anti-cancer mechanisms of clinically acceptable colchicine concentrations on hepatocellular carcinoma. Life Sci. 2013 Sep 3;93(8):323-8. doi: 10.1016/j.lfs.2013.07.002. Epub 2013 Jul 16. PMID 23871804
- [Background] Wu CC, Lin ZY, Kuoc CH, Chuang WL. Clinically acceptable colchicine concentrations have potential for the palliative treatment of human cholangiocarcinoma. Kaohsiung J Med Sci. 2015 May;31(5):229-34. doi: 10.1016/j.kjms.2015.01.008. Epub 2015 Mar 10. PMID 25910557
- [Background] Lin ZY, Kuo CH, Wu DC, Chuang WL. Anticancer effects of clinically acceptable colchicine concentrations on human gastric cancer cell lines. Kaohsiung J Med Sci. 2016 Feb;32(2):68-73. doi: 10.1016/j.kjms.2015.12.006. Epub 2016 Feb 2. PMID 26944324
- [Derived] Lin ZY, Yeh ML, Liang PC, Chen SC, Huang CF, Huang JF, Dai CY, Yu ML, Chuang WL. Phase IIb Trial for the Palliative Treatment of Patients With Primary Hepatic Malignancy Unable to Receive Curative Treatment: Efficacy of Colchicine. Kaohsiung J Med Sci. 2025 Sep 27:e70121. doi: 10.1002/kjm2.70121. Online ahead of print. PMID 41014140